CLINICAL TRIAL: NCT07092332
Title: Young Vulvodynia: Effect and Efficacy of a Multimodal Treatment for Young Women With Vulvar Pain
Brief Title: Young Vulvodynia: Effect and Efficacy of Multimodal Treatment.
Acronym: UV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Rebecca Lennartsson, Doctoral Student, Region Örebro County
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 282171; RFR-1010966 (Other Grant/Funding Number: Regional Research Council Mid Sweden); OLL-1013529 (Other Grant/Funding Number: Nyckelfonden)
Record Dates: First submitted 2025-06-10; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Vulvodynia
Keywords: Vulvodynia; Provoked Vulvodynia; Multimodal Treatment; Cognitive Behavior Therapy; Single-Case Experimental Design; Chronic Pain; Adolescent; Emerging Adulthood
MeSH Terms: conditions — Vulvodynia; Chronic Pain | interventions — Combined Modality Therapy

STUDY DESIGN:
Intervention Model Description: The study utilises a sequential single-case experimental AB design with randomized waiting period length (4, 5 or 6 weeks). Included in the design is also a pre-, post- and 6 month follow up measurement allowing for single group analysis of change. In addition, we collect qualitative data from patients, to explore experiences of participation in the study and the treatment.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to baseline length allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baseline period (No Intervention): During a 4, 5 or 6 week waiting period, participants respond to a short questionnaire twice a week.
- Multimodal Treatment (Experimental): Multimodal Treatment.
  Interventions: Behavioral: Multimodal treatment

INTERVENTIONS:
Behavioral: Multimodal treatment — Vulvodynia Intervention adapted for late adolescents and young adults. A multimodal treatment for provoked vulvodynia
  The treatment consists of 11 treatment sessions. Working with goal-directed behavior change that has both physiological and psychosocial components. The treatment sessions will be conducted with various professionals, bot simultaneously and separately.
  The intervention is based on physiological and psychosocial components working with goal-directed behavioral change; both educational and practical elements, examples of these are vulva care, lubrication exercises, pelvic floor relaxation, work with thoughts, feelings, and behaviors related to the pain, as well as thoughts, feelings and behaviors related to sex and desire, and educational and practical elements focusing on open communication and validation. The treatment sessions are between 60 to 90 minutes each. There is a possibility for the participants to involve partner during two of the treatment sessions.
  Arms: Multimodal Treatment

SUMMARY:
The aim of this SCED-study is to evaluate a multimodal treatment for vulvodynia in young women. The main questions it aims to answer are:

Is multimodal treatment effective for provoked vulvodynia in young women? How is multimodal treatment experienced by young women with vulvodynia?

Participants will respond to frequent questionnaires (two times a week) during a baseline period of 4,5 or 6 weeks, as well as during their treatment period ( a total of 25 weeks). In addition they will respond to pre-, post-treatment and 6 month follow-up questionnaires.

DETAILED DESCRIPTION:
The current study is an effectiveness evaluation, applying a sequential single case experimental AB design (SCED) with randomized baseline length, implemented at a youth guidance center. Potential participants will be informed about the study and answer a few questions digitally to ensure that participation in the study is appropriate for them. An assessment will then be conducted and questions will be asked about the pain, psychological, sexual and relational health, and a diagnostic interview will be conducted to exclude other psychological issues that needs to be prioritized before vulvodynia treatment.

After the assessment interview and inclusion, participants will be randomized in tiers to a 4, 5, or 6 week baseline period. Thereafter, the treatment will begin. During the baseline and treatment period, participants will complete a short self-assessment questionnaire, twice a week, to measure pain (primary outcome) and other key variables. To facilitate the repeated assessments, we will use the m-Path app, which was developed by KU Leuven University in Belgium to easily evaluate treatment for both patients and therapists. In addition to the repeated assessments, the treatment will be evaluated through a comprehensive web-based self-assessment questionnaire before and after the intervention and at a six-month follow-up. The outcome measures are in line with Core Outcome set in Vulvodynia.

ELIGIBILITY:
Inclusion Criteria:

* Biological sex female
* 15-23 years of age
* Diagnosed with Provoked vulvodynia

Exclusion Criteria:

* Severe psychological issues that should be prioritized before vulvodynia treatment (e.g., substance abuse, psychosis)
* Ongoing pregnancy
* Childbirth within the last year
* Post-traumatic stress disorder (PTSD) related to sexual trauma
* Insufficient mastery of the Swedish language
* No experience of vaginal sex, as vaginismus might be suspected, which requires different treatment

Ages: 15 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Genital Pain Intensity | Pre, post treatment (25 weeks after the baseline measurement started) and at 6 month follow-up. Repeated measures twice a week during baseline (4, 5 or 6 weeks) and treatment period, for 25 weeks.
  Provoked pain during sexual and non-sexual activities. Seven activities where pain is rated on a scale from 0 to 10. Higher scoring indicates higher degree of pain. There are also subsequent questions regarding whether they have performed the described activity or not within a specific time frame.

SECONDARY OUTCOMES:
Sexual Function | FSFI: Pre, post treatment (25 weeks after the baseline measurement started) and at 6 month follow-up. FSFI-6 Repeated measures twice a week during baseline (4, 5 or 6 weeks) and treatment period, for 25 weeks.
  The Female Sexual Function Index (FSFI) is a self-report measure of female sexual function that assesses six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. It consists of 19 questions, rated on a 5-point scale, with a higher score indicating a better sexual function. The short version, FSFI-6 contains 6 questions.
Participant Identified Treatment Goal | Pre, post treatment (25 weeks after the baseline measurement started) and at 6 month follow-up. Repeated measures twice a week during baseline (4, 5 or 6 weeks) and treatment period, for 25 weeks.
  All participants identify one own primary goal. Participants chose an individual treatment goal and rate treatment goal attainment, from 0-10, 0= the goal is not at all achieved, 10= the goal is achieved.
Pelvic Floor Tension | Pre, post treatment (25 weeks after the baseline measurement started) and at a 6 month follow-up. During baseline and treatment period measured twice a week, for 25 weeks.
  Self-report assessment of pelvic floor tension and pelvic floor relaxation. Two items rated on a 11-point scale, from 0-10, higher scores indicate greater tension and more difficulty relaxing the pelvic floor, and physiotherapeutic examination.
Sexual Satisfaction | Pre and post treatment (25 weeks after the baseline measurement started) and at 6 months follow-up
  Sexual Satisfaction as measured with Global Measure of Sexual Satisfaction (GMSEX), 5 items rated on a 7 point scale. Higher scores indicate a higher degree of sexual function.
Sexual Pain Coping | Pre, post treatment (25 weeks after the baseline measurement started) and at 6 month follow-up, during baseline (4, 5 or 6 weeks) and treatment period measured twice a week for 25 weeks´.
  Avoidance and Endurance Coping strategies related to sexual pain. Measured with CHAMP Sexual Pain Coping Scale. 12 items assess coping strategies for sexual pain: avoidance and endurance, rated on a 7 point-scale from 1 to 7, where higher scoring indicating a higher degree of avoidance and/or endurance.
  For repeated measure: Two items from the CHAMP Sexual Pain Coping Scale (CSPCS), rated on a 7-point scale, with higher scores indicating a higher degree of avoidance and endurance.
Pain Catastrophizing | Pre and post treatment (25 weeks after the baseline measurement started) and at 6 months follow-up
  Pain Catastrophizing, as measured by the CSQ-CAT. 7 items rated on a 5-point scale from 0 (not at all) to 4 (all the time). Higher scores indicating greater levels of pain catastrophizing.
Depressive symptoms | Pre and post treatment, and at 6 months follow-up
  Using the patient health questionnaire (PHQ-9), 9 items are rated on a 4-point scale, from 0 to 3. Higher scores indicating higher degree of depression symtoms.
Anxiety symptoms | Pre- and post treatment and at 6 month follow-up.
  Using the Generalized Anxiety Disorder questionnaire (GAD-7), 7 items rated on a 4-point scale from 0 to 3, higher scoring indicating a higher degree of anxiety symptoms.
Change in quality of life | Pre and post treatment, and at 6 months follow-up
  World Health Organization Quality of Life-BREF, 1 item where participants rates their quality of life, on a 5-point scale from 1 to 5, higher scoring indicating greater quality of life.
Change in life interference, sexual function interference and communication. | Pre and post treatment (25 weeks after the baseline measurement started) and at 6 months follow-up
  Vulvar pain assessment questionnaire (VPAQ)-short Inventory is a disease-specific set of measurement scales to capture the biopsychosocial nature of vulvodynia. We are using the parts from the questionnaire that evaluates life interference, sexual function interference, impact on relationship and sexual communication.
  Life interference:6 items rated on a 6-point scale from 0 (not at all) to 4 (avoid because of pain). Higher scores indicating greater life interference.
  Sexual function interference: 5 items rated on a 6-point scale from 0 (not at all) to 4 (avoid because of pain)
  6 items about communication with partner rated on a 5-point scale from 0 (largely uncomfortable) to 4 (largely comfortable). Higher scoring indicates

OTHER OUTCOMES:
Demographic | Pre treatment. Questions about partner/-s are measured pre and post treatment and at 6 month follow-up.
  Age, country of birth, educational level, occupation, if they have a partner/-s, how long they have been in that relationship/-s, gender of partner/-s, if they have kids, childbirth during the last year, ongoing pregnancy, menstruation
Experiences of sexual and physical abuse | Pre-treatment
  Using the Sexual and Physical Abuse Questionnaire (SPAQ).
Treatment expectations | Pre-treatment
  2 items rated on a 11-point scale, from 0 to 10. Higher scoring indicating higher expectations that this treatment will be helpful.
Negative treatment effects | Post-treatment
  1-2 items measuring negative effects of the treatment. One questions that asks if the participant experienced any negative effects of the treatment, with a following question asking the participant to describe more in an open answer.
Perceived treatment improvement and satisfaction | Post treatment
  4 items rating potential improvement and satisfaction on a 6-point scale (1-6), higher scoring indicating greater improvement and satisfaction
Experience of treatment | Post-treatment
  Semi structured interviews, individual interviews and focus groups, probing qualitative aspects of the treatment experience, and the experience of implementation of patients, treating practitioners and clinical managers.

CONTACTS AND LOCATIONS:
Locations (1):
- Ungdomsmottagningen, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No
Because of the sensitive nature of the data. Data can be provided by request.